CLINICAL TRIAL: NCT05250440
Title: Noninvasive and Dynamic Monitoring the Biological Parameters of Eyes in Different Age Groups
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022020901
Record Dates: First submitted 2022-02-10; First posted 2022-02-22 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2022-02

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- (a1)Emmetropia: +0.75 to -0.75 D: age: 12 to 18 years old
- (a2)Mild myopia: -1.00 to -3.00 D: age: 12 to 18 years old
- (a3)Moderate myopia: -3.25 to -6.00 D: age: 12 to 18 years old
- (a4)High myopia: >-6.00 D: age: 12 to 18 years old
- (b1)Emmetropia: +0.75 to -0.75 D: age: 18 to 35 years old
- (b2)Mild myopia: -1.00 to -3.00 D: age: 18 to 35 years old
- (b3)Moderate myopia: -3.25 to -6.00 D: age: 18 to 35 years old
- (b4)High myopia: >-6.00 D: age: 18 to 35 years old

SUMMARY:
Myopia is the most common refractive eye disease worldwide. The number of cases is up to 2 billion. In recent years, the incidence of myopia in China is obviously rising trend. As early as the 2018 national health committee epidemiological data show that teenage myopia rate in China has been the first in the world, and has become the influence in China, especially the youth eye health major public health problem. In recent years, prevention and control measures for myopia have emerged in endlessly, such as increasing outdoor activity time, sufficient sunlight exposure, orthokeratology and local use of low-concentration atropine can partially prevent the occurrence or slow down the progression of myopia. But the effects are limited and cannot completely inhibit the development of myopia.

In recent years, with the in-depth study of myopia, it is found that myopia is not only the change of diopter, but also the pathological changes of the whole eyeball shape and corresponding tissues. The incidence of myopia is closely related to the biological parameters of the eyeball, which has become a hotspot of clinical research in recent years. Current studies believe that eyeball biological parameters such as axial length, scleral thickness, choroid thickness are related to the occurrence of myopia, among which the change of scleral structure and shape, namely scleral remodeling, is considered to be an important factor in all visual stimuli leading to myopia. A large number of studies have also shown that scleral remodeling can lead to changes in the scleral biomechanics, thereby promoting the development of myopia. Multiple studies have shown a negative correlation between myopia and scleral thickness, with the thinning of the lower anterior sclera being the most significant. The lower anterior sclera is considered to be a marker for predicting the development of myopia, but some studies have found no correlation between the two. Such differences in the results may be related to the precision of the measurement instrument, the sample size of the included cases, age, and the grouping of different refractive states. The correlation between various biological parameters of the eyeball, especially the sclera, and myopia is not clear at present. Therefore, more penetrating and clearer instruments, more sample sizes, and more scientific grouping are needed for further research and confirmation.

DETAILED DESCRIPTION:
The Department of Ophthalmology, Zhongnan Hospital of Wuhan University, has a variety of the most advanced instruments and equipment in the world, such as the newly listed TOMEY CASIA2, which is non-invasive and non-contact, and can quickly obtain the living body tomography of the anterior part of the eye tissue structure at one time, and can conduct quantitative analysis. The latest generation of Ultra Wide Angle fundus imager (Optoc) that is, under the small pupil to obtain nearly 200 degrees fundus image, Heidelberg confocal fundus diagnostic instrument, IOL MASTER700 biometric instrument, etc. This topic is proposed to use an eye the forefront of the latest generation of instruments and equipment, to emmetropia, mild myopia, moderate myopia and high myopia eyeball all biological parameters measurement, explore various biological parameters and the correlation of myopia, for myopia prevention and control such as nearsightedness in the process of the follow-up biological indicators need to focus on monitoring, provide powerful clinical basis.

ELIGIBILITY:
Inclusion Criteria:

* Resident population in Hubei Province
* No gender preference
* Healthy population aged between 12 and 35

Exclusion Criteria:

* Systemic diseases
* History of other eye diseases, surgery and/or medications, and eye trauma
* Anisometropia > 2.00 D
* Astigmatism > 2.00 D
* The best corrected visual acuity was less than 0.8

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 1. Resident population in Hubei Province
  2. No gender preference
  3. Healthy population aged between 12 and 35
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Axial length | 10 am to 12 am, every day
  Axial length was measured by IOL Master700 partially coherent interferometry.
Anterior scleral thickness | 10 am to 12 am, every day
  Anterior segment OCT images used to determine anterior scleral thickness obtained by gazing in 4 directions (superior, temporal, inferior, and nasal).
Posterior scleral thickness | 10 am to 12 am, every day
  Spectralis HRA+OCT images used to determine posterior scleral thickness under fovea.
Choroid thickness | 10 am to 12 am, every day
  Spectralis HRA+OCT images used to determine choroid thickness obtained by gazing in 4 directions (superior, temporal, inferior, and nasal).

CONTACTS AND LOCATIONS:
Overall Officials: Min Ke, Doctor, Study Director — Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided
gender, age, refractive diopter, best corrected visual acuity, ocular axial length, anterior scleral thickness, choroid thickness, posterior scleral thickness